CLINICAL TRIAL: NCT03533530
Title: Electrical Source Imaging in Presurgical Evaluation of Patients With Focal Epilepsy: A Prospective Study of Clinical Utility
Brief Title: Clinical Utility of ESI in Presurgical Evaluation of Patients With Epilepsy
Acronym: CUESIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Filadelfia Epilepsy Hospital (Other); Lundbeck Foundation (Other); Lennart Grams Mindefond, Danish Epilepsy Society (Unknown)
Responsible Party: Principal Investigator, Olaf B Paulson, Professor, MD, DMSc, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: LD&HD-ESI
Record Dates: First submitted 2018-04-26; First posted 2018-05-23 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Electroencephalography; Refractory Epilepsy; Brain Imaging; Surgery
Keywords: Electrical source imaging
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: Evaluation of low-density (LD, 25 channels) and high-density (HD, 256 channels) electrical source imaging (ESI) in epilepsy surgery
Who Masked: Outcomes Assessor
Masking Description: The Epilepsy Surgery Group make their decision about the surgical approach only with knowledge of the LD-EEG without ESI (and knowledge of non EEG investigations). Thereafter the LD ESI results are revealed and the clinical decision is revised. Finally the HD ESI results are revealed and the clinical decision is revised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No electrical source imaging (ESI) (Active Comparator): In all patients, the multidisciplinary epilepsy surgery team will make a conclusion on management plan, based on all non-invasive presurgical data, except for ESI.
  Interventions: Diagnostic Test: No electrical source imaging (ESI)
- Low-density ESI (LD ESI) (Experimental): The multidisciplinary epilepsy surgery team will make a conclusion on management plan, based on all non-invasive presurgical data, including ESI using LD EEG recordings.
  Interventions: Diagnostic Test: Low-density ESI (LD ESI)
- High-density ESI (HD ESI) (Experimental): The multidisciplinary epilepsy surgery team will make a conclusion on management plan, based on all non-invasive presurgical data, including ESI using HD EEG recordings.
  Interventions: Diagnostic Test: High-density ESI (HD ESI)

INTERVENTIONS:
Diagnostic Test: Low-density ESI (LD ESI) — Electrical source imaging using low density EEG
  Arms: Low-density ESI (LD ESI)
Diagnostic Test: High-density ESI (HD ESI) — Electrical source imaging using high density EEG
  Arms: High-density ESI (HD ESI)
Diagnostic Test: No electrical source imaging (ESI) — For all patients: MRI, semiology, visual interpretation of EEG. When needed: PET, SPECT.
  Arms: No electrical source imaging (ESI)

SUMMARY:
This study evaluates to what extend electrical source imaging (ESI) provides nonredundant information in the evaluation of epilepsy surgery candidates. Epilepsy surgery normally requires an extensive multimodal workup to identify the epileptic focus. This workup includes Magnetic Resonance Imaging (MRI), electroencephalography (EEG) without source imaging, video monitoring and when needed Positron Emission Tomography (PET), Magnetoencephalography (MEG), Single Photon Emission Computed Tomography (SPECT) and invasive EEG recordings using implanted electrodes. ESI estimates the location of the epileptic source with a high sensitivity and specificity using inverse source estimation methods on non-invasive EEG recordings. This study aims to investigate the clinical utility of ESI using low-density (LD, 25 channels) and high-density (HD, 256 channels) EEG. Clinical utility is defined in this study as the proportion of patients in whom the patient management plan was changed, based on the results of ESI. Should ESI be added to the routine work-up of epilepsy surgery candidates.

DETAILED DESCRIPTION:
Patients with drug resistant epilepsy can be offered resective neurosurgery if seizure semiology, video-EEG and MRI points to a focal origin in the brain. Are these investigations not concordant or is the MRI without a lesion, then additional investigations such as PET, SPECT and MEG can be performed before deciding upon operation or further, invasive investigation, using intracranial EEG recordings. If a single hypothesis can be made the patient can be operated. In case of one main hypothesis and additional hypothesis, intracranial EEG registration can be performed. If there are no hypothesis or too many hypotheses the patient cannot be offered surgery.

In the present study electrical source imaging (ESI) will be performed in epilepsy surgery candidates on low density (LD, 25 channels) and high density (HD, 256 channels) electroencephalography (EEG). In the analysis of LD-EEG, a template brain and template electrode position will be used. In the analysis of HD-EEG an individual MRI scan and individual electrode position will be used.

The multidisciplinary epilepsy surgery team will be blinded to the results of the ESI, until based on MRI, LD EEG (without source imaging), video monitoring and optionally PET, MEG and ictal-SPECT, the investigators have decided whether a patient 1) is ready for surgery, 2) should be evaluated with intracranial electrodes or 3) cannot be offered operation. This decision is registered. Then LD ESI is presented. It is registered whether any change in the patient management plan was made, based on the ESI data. Further, for 1) it is registered whether the planned extend of the surgical resection is changed and whether intraoperative EEG recording is needed; for 2) it is registered if the planned implantation strategy of intracranial electrodes is changed; and for 3) whether other additional evaluation is needed. Finally, HD ESI is presented and it is registered if this changes the decision made without ESI, according to the above-mentioned categories.

Clinical utility of LD ESI and of HD ESI is defined as the proportion of patients in whom the patient management plan was changed, based on the LD ESI and respectively HD ESI. The investigators will use McNemar test to compare the proportion of changes based on LD ESI with those based on HD ESI. The localization provided by the ESI methods, will be compared with the conclusion of the multidisciplinary team, on the localization of the epileptic focus. In patients having intracranial EEG performed within the study period, the results will be compared to the ESI results. In patients having one-year follow-up after operation and being seizure free, it will be evaluated if the location of the ESI was within the operation area.

ELIGIBILITY:
Inclusion Criteria:

* Drug resistant epilepsy
* Potential candidates for epilepsy surgery

Exclusion Criteria:

* Can not cooperate for EEG recording

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Clinical utility of LD ESI and of HD ESI: change in clinical decision following ESI | Through study completion - an average 1 year - at the end of the presurgical work-up of each patient, at the multidisciplinary epilepsy surgery meeting. The timeframe of completing the presurgical evaluation varies from 6 months to 24 month.
  Defined as the proportion of patients in whom the patient management plan was changed, based on the LD ESI and respectively HD ESI

SECONDARY OUTCOMES:
Change to stop | Through study completion - an average 1 year - at the end of the presurgical work-up of each patient, at the multidisciplinary epilepsy surgery meeting. The timeframe of completing the presurgical evaluation varies from 6 months to 24 month.
  The patient is not offered surgery.
Change from stop to implantation of intracranial electrodes | Through study completion - an average 1 year - at the end of the presurgical work-up of each patient, at the multidisciplinary epilepsy surgery meeting. The timeframe of completing the presurgical evaluation varies from 6 months to 24 month.
  Without ESI the patient is not offered surgery. Based on ESI, implantation of intracranial recordings is offered.
Change in the strategy (location) of implanted intracranial electrodes | Through study completion - an average 1 year - at the end of the presurgical work-up of each patient, at the multidisciplinary epilepsy surgery meeting. The timeframe of completing the presurgical evaluation varies from 6 months to 24 month.
  Additional intracranial electrodes are implanted, based on the results of ESI.
Change from stop to operation | Through study completion - an average 1 year - at the end of the presurgical work-up of each patient, at the multidisciplinary epilepsy surgery meeting. The timeframe of completing the presurgical evaluation varies from 6 months to 24 month.
  Without ESI, the patient is not offered operation. Based on ESI, operation is offered.
Change from implantation of intracranial electrodes to operation | Through study completion - an average 1 year - at the end of the presurgical work-up of each patient, at the multidisciplinary epilepsy surgery meeting. The timeframe of completing the presurgical evaluation varies from 6 months to 24 month.
  Without ESI, implantation of intracranial electrodes is offered. Based on ESI, operation is offered.
Change from operation to implantation of intracranial electrodes | Through study completion - an average 1 year - at the end of the presurgical work-up of each patient, at the multidisciplinary epilepsy surgery meeting. The timeframe of completing the presurgical evaluation varies from 6 months to 24 month.
  Without ESI, operation is offered. Based on ESI this is changed to implantation of intracranial electrodes.

OTHER OUTCOMES:
The localization provided by the ESI methods, will be compared with results of the intracranial recordings and the operation outcome (where available) | An average 1 year - at follow-up of the intracranial results and following the operation. The timeframe for follow-up varies from 6 months to 18 month.
  Comparison at sublobar level between the ESI and the conclusion of the multidisciplinary team.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf B Paulson, MD, DMSc, Principal Investigator — Rigshospitalet, N-6931
Locations (1):
- Rigshospitalet, Copenhagen, Select, Denmark

IPD SHARING:
Plan to Share IPD: No